CLINICAL TRIAL: NCT02524925
Title: Postoperative Stress Response in Patients Following Fast Track Versus Conventional Protocol After Hepatectomy or Pancreatectomy
Brief Title: Postoperative Stress Response in Patients Following Fast Track vs Conventional Protocol After Hepatectomy or Pancreatectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Collaborators: Saint Savvas Anticancer Hospital (Other)
Responsible Party: Principal Investigator, Maria Kapritsou, RN, BSc, MSc, PhD(c), National and Kapodistrian University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 87
Record Dates: First submitted 2015-08-10; First posted 2015-08-17 (Estimated); Last update posted 2015-08-17 (Estimated); Status verified 2015-08

CONDITIONS: Hepatic Cancer; Cancer of Pancreas
Keywords: fast track surgery; eras program; hepatectomy; pancreatectomy; NPY; ACTH/Cortsiosol; postoperative stress
MeSH Terms: conditions — Liver Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- fast track protocol (Active Comparator): Oral fluids intake (0.5 lt) 6 hours after operation Mobilization 4 hours after operation Check discharge criteria the 4th-6th postoperative day
  Interventions: Procedure: fast track protocol
- conventional protocol (No Intervention): Oral intake after bowel mobilization Mobilization after the 1st postoperative day Check discharge criteria the 7th-15th postoperative day

INTERVENTIONS:
Procedure: fast track protocol — Evaluation of postoperative stress
  Arms: fast track protocol

SUMMARY:
A prospective randomized clinical study, with cross-sectional comparisons and correlations was conducted from May 2012 to July 2015 with a sample of 231 patients who have undergone hepatectomy or pancreatectomy, randomized into 2 groups. In group A was applied postoperatively the protocol Fast-track, while in group B the conventional postoperative care. Demographic and clinical data were collected. In 170 patients, Neuropeptide Y (NPY), Adrenocorticotropic hormone (ACTH)/Cortisol plasma levels were measured by ELISA method: a) at the day of patient's admission, b) the operation day, c) the 3rd postoperative day or prior to discharge.

DETAILED DESCRIPTION:
Pain levels were assessed by Puntillo scale (behavioral observation scale) which has ranges; 0-1 "no pain", 2-4 "aching" 5-7 "moderate pain" 8-10 and "severe pain".

Patient stress levels were evaluated by: a) scale I.C.U.E.S.S. which evaluated environmental stress during their stay in hospital and takes values; 40-80 "no environmental stress" 81-120 "mild to moderate environmental stress," 121-160 " Moderate to severe environmental stress ", b) three questions of self- experienced feelings (with a score of 0 = None and 10 = Completely) like "How sad you feel right now?" "How stress do you feel right now?" "How optimist do you feel right now about the future?" The data collected in three phases: a) the day of hospitalization, b) the day of surgery, and c) the third postoperative day or before discharge.

Depression levels were evaluated with Zung scale (Zung self-rating depression scale), which assesses depression levels with a score 25-49 for "normal level mood," 50-59 for "mild depression", 60-69 for "moderate depression" and 70 + for "severe depression".

ELIGIBILITY:
Inclusion Criteria:

* patients with American Society of Anesthesiologists (ASA) PHYSICAL STATUS CLASSIFICATION SYSTEM I-III
* age 30-82 years,
* with normal level of consciousness and communication

Exclusion Criteria:

* the presence of chronic pain,
* kidney disease, neuropathy,
* systemic as well as chronic treatment with analgesics

Ages: 30 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 231 (Actual)
Dates: Start 2012-04; Primary Completion 2015-03 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Analyzing Neuropeptide Y, Cortisol and Adrenocorticotropic hormones levels in blood samples | Participants will be followed for the duration of hospital stay, an expected average of 15 days
  Analyzing Neuropeptide Y, Cortisol and Adrenocorticotropic hormones levels in blood samples in patients after hepatectomy or pancreatectomy. These measures will occured in three phases a. the day of hospitalzation, b. the day of surgery c. the day of discharge.

SECONDARY OUTCOMES:
Evaluating postoporative stress between the two protocols with scales | Participants will be followed for the duration of hospital stay, an expected average of 15 days
  Evaluating postoporative stress with scales, such as Zung scale the day of hospitalization, ICUESS scale the 3rd postoperative day, Puntillo scale the day of surgery and three self-experienced questions how sad are you feeling, how stressed are you feeling and how optimistic are you feeling in three phases:a. the day of hospitalzation, b. the day of surgery c. the day of discharge.
Evaluating postoperative pain between the two protocols with scale | Participants will be followed for the duration of hospital stay, an expected average of 15 days
  Evaluating postoperative pain between the two protocols with scale such as Puntillo scale the day of surgery

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos A Konstantinou, RN, PhD, Study Director — National and Kapodistrian University of Athens